CLINICAL TRIAL: NCT00573911
Title: Acid Reflux and Stromal Fibroblasts in Barrett's Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Prasad G. Iyer, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-002453; IRUSESOM0546
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Barrett's Esophagus; GERD
Keywords: Barrett's esophagus; GERD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Endoscopy and pH study — endoscopy and PH study done one time

SUMMARY:
Patients with Barrett's Esophagus are known to have excessive distal esophageal acid exposure comparable to patients with erosive esophagitis. A significant proportion of patients with BE who are not symptomatic on treatment continue to have persistent acid reflux. High dose esomeprazole is able to control acid reflux in patients with BE. The effect of acid reflux on Barrett's esophagus stroma is currently unknown.

It is our hypothesis that stromal fibroblast activation in Barrett's esophagus is influenced by acid reflux. The specific aim of this proposal will be: To assess the association between acid reflux and subepithelial fibroblasts in Barrett's esophagus.

DETAILED DESCRIPTION:
We will conduct a prospective cohort study to assess the degree of stromal activation in patients with LSBE (without dysplasia) who have adequate and inadequate control of acid reflux in the distal esophagus. The study will be conducted in two phases.

Phase 1 (Pilot): 20 patients with LSBE without dysplasia will undergo endoscopy with biopsies and a 24 hour pH study on treatment. Patients will then be divided into 2 groups:

* Group A (GER): Those with ongoing acid reflux (characterized by either presence of esophagitis [LA classification B,C or D1] on endoscopy, and/or a positive pH study on treatment defined using standard criteria)
* Group B (NGER): Those with controlled acid reflux (negative endoscopy and pH study on treatment).

Stromal markers that will be assessed and compared between the 2 groups will include: presence of activated myofibroblasts (detected by immunohistochemistry for vimentin and smooth muscle actin).

ELIGIBILITY:
Inclusion Criteria:

* Prior histological demonstration of Barrett's esophagus that is endoscopically visible; length of visible segment >/= 1 cms
* Absence of dysplasia on prior biopsies
* Laboratory studies:

  * Prothrombin time (INR) < 1.5
  * Hemoglobin > 8.0 gm/dL
* Ability to provide informed consent

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status 3 or 4
* Inability to tolerate endoscopic procedures
* Pregnancy: Females of child-bearing age will be screened with pregnancy test. Although none of the procedures in the study are contraindicated in pregnancy, sedation used in endoscopy can be contraindicated in early pregnancy
* Prior esophageal surgery, or cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The specific aim of this proposal will be: To assess the association between acid reflux and subepithelial fibroblasts in Barrett's esophagus. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States